CLINICAL TRIAL: NCT06000930
Title: Cardiac Troponin Fragmentation After Heavy Physical Exercise The MaraCat2 Study
Acronym: MaraCat2
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, University of Turku
Other Study IDs: 13.06.2023/207
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction; Myocardial Injury
Keywords: exercise; troponin; myocardial infarction; myocardial injury
MeSH Terms: conditions — Myocardial Infarction; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- marathon runners: Marathon runners
  Interventions: Diagnostic Test: Troponin fragmentation
- myocardial infarction: Patients with Type 1 myocardial infarction
  Interventions: Diagnostic Test: Troponin fragmentation

INTERVENTIONS:
Diagnostic Test: Troponin fragmentation — laboratory test from blood sample

SUMMARY:
Cardiac troponins are highly sensitive and specific biomarkers of cardiac injury and are in a key role in the diagnosis of acute myocardial infarction (MI). Minor troponin elevations are common after prolonged strenuous exercise without clinical symptoms of MI or myocardial injury. Importantly, currently used high-sensitivity troponin T (cTnT) test detects also smaller troponin fragments which may cause troponin elevation after exercise and lead to false diagnosis of MI.

In the present study protocol, we compare the characteristics troponin release after marathon race and Type 1 MI with the improved version of our novel troponin fragmentation test (SuperTropo test) and the commercial cTnT test.

A total of 65 recreational runners participating in the 2023 Paavo Nurmi Marathon in Turku are recruited. All participants give a blood sample during the post-race visit (within 30 min after finishing the marathon).

A control group of 90 patients with acute Type 1 MI are recruited among patients admitted to Heart Centre of Turku University Hospital.

Commercial cTnT and long troponin component of cTnT analyzed witha novel immunoassay are dtermined in all subjects to assess cTnT fragmentation. TYhe main aims of the study are:

To assess how often cTnT is elevated after marathon running and which factors affect the cTnT rise? Is the fragmentation of troponin more common after marathon race compared with Type 1 MI and can the novel Supertropo test separate execise-induced troponin rise from those caused by MI ?

DETAILED DESCRIPTION:
Cardiac troponins are highly sensitive and specific biomarkers of cardiac injury and are in a key role in the diagnosis of acute myocardial infarction (MI). Minor troponin elevations are common after prolonged strenuous exercise without clinical symptoms of MI or myocardial injury.

Based on a small gel filtration chromatography study the released troponin in this condition seems to be predominantly in the form of small fragments. These smaller cytosolic troponin fragments may more easily traverse across cell membranes that have become leaky but not irreversibly damaged. Importantly, currently used high-sensitivity troponin T (cTnT) test detects also smaller troponin fragments which may lead to false diagnosis of MI.

In a Proof-of-Principle study we developed a novel immunoassay which is much simpler and more sensitive than previously used laboratory methods for studying cTnT fragmentation. In the present study protocol, we compare the characteristics troponin release after marathon race and Type 1 MI with the improved version of our novel troponin fragmentation test (SuperTropo test) and the commercial cTnT test.

A total of 65 recreational runners participating in the 2023 Paavo Nurmi Marathon in Turku are recruited to the MaraCat2 Study with an open email invitation. All participants give a blood sample during the post-race visit (within 60 min after finishing the marathon).

A control group of 90 patients with acute Type 1 MI are recruited among patients admitted to Heart Centre of Turku University Hospital. Coronary angiography is performed in all included patients to confirm culprit lesion and the MI diagnosis. All included patients are treated with primary or urgent percutaneous coronary intervention. Only patients with <24 delay from symptom onset to blood sample are included to avoid the effects of later gradual fragmentation of cTnT in the circulation.

Certified laboratory services by Turku University Hospital (TYKSLAB) take care of blood samples. After centrifugation, serum is aliquoted, frozen and stored at -70 °C for later analysis. Analysis is performed on a single day using the same calibration and set-up to minimize variation.

cTnT was analyzed using a commercial high-sensitive assay (Roche Diagnostics GmbH, Mannheim, Germany).

A novel sensitive time-resolved immunofluorometric assay is used for the detection of long cTnT forms (long cTnT). The long cTnT assay follows the sandwich type immunoassay format and utilizes time-resolved-fluorescence (TRF) as the measurement platform.

The main aims of the study are:

To assess how often cTnT is elevated after marathon running and which factors affect the cTnT rise? Is the fragmentation of troponin complex (assessed by long cTnT/ total cTnT ratio) more common after marathon race compared with Type 1 MI? Is the novel Supertropo test able to separate exercise-induced troponin elevations from those caused by MI ? All participants provide written informed consent. The study complies with Declaration of Helsinki as revised in 2002 and the study protocol was approved by the Medical Ethics Committee of the Hospital District of Southwest Finland.

Statistical analysis Continuous variables are reported as mean ± standard deviation when normally distributed, and as median [inter-quartile range (IQR)] if they were skewed unless stated otherwise. The normality of the data distribution is examined by the Shapiro-Wilk test. Statistical significance was assumed at a p value < 0.05. Categorical variables were described with absolute and relative (percentage) frequencies. Chi-squared test and Fisher's exact test are used for categorical variables as appropriate. Independent samples t-test and Mann-Whitney U test are used for univariate analysis. Correlation between continuous variables are estimated using the Spearman test. Linear regression analysis with backward selection is used to identify factors significantly relating to post-race cTnT levels. All predictors with a P value < 0.1 in univariate analysis were included in the final regression model.

ELIGIBILITY:
Inclusion Criteria:

* participating marathon race or treated for Type 1 myocardial infarction and giving informed consent

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Marathon runners and patients with acute myocardial infarction as a control group
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-08-19 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Magnitude of Troponin fragmentation in the post-race and post-MI (<24h) blood samples | < 1 hour after marathon race and < 24 hours after myocardial infarction
  Ratio of long troponin component to total troponin T in the post-race and post-MI (<24h) blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Juhani K Airaksinen, Md, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Airaksinen KEJ, Paana T, Vasankari T, Salonen S, Tuominen T, Linko-Parvinen A, Pallari HM, Hellman T, Teppo K, Heinonen OJ, Jaakkola S, Wittfooth S. Composition of cardiac troponin release differs after marathon running and myocardial infarction. Open Heart. 2024 Nov 17;11(2):e002954. doi: 10.1136/openhrt-2024-002954. PMID 39551608